CLINICAL TRIAL: NCT02740712
Title: A Phase 1, Open-label, Multiple-probe Drug-drug Interaction Study to Determine the Effect of Rucaparib on Pharmacokinetics of Caffeine, S-Warfarin, Omeprazole, Midazolam, and Digoxin in Patients With Advanced Solid Tumors
Brief Title: Pharmacokinetic Drug-Drug Interaction Study of Rucaparib
Acronym: DDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: pharmaand GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CO-338-044
Record Dates: First submitted 2016-03-30; First posted 2016-04-15 (Estimated); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Neoplasms
Keywords: rucaparib; CO-338; Clovis; Clovis Oncology; PARP Inhibitor; Drug-Drug Interaction
MeSH Terms: conditions — Neoplasms | interventions — Caffeine; Warfarin; Omeprazole; major urinary proteins; Midazolam; Digoxin; Vitamin K; rucaparib

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm probe drugs and rucaparib (Other): Caffeine Warfarin Vitamin K Omeprazole Midazolam Digoxin rucaparib
  Interventions: Drug: Caffeine; Drug: Warfarin; Drug: Omeprazole; Drug: Midazolam; Drug: digoxin; Drug: Vitamin K; Drug: Rucaparib

INTERVENTIONS:
Drug: Caffeine — 200 mg (4 x 50mg) Tablet
Drug: Warfarin — 10 mg (2 x 5mg) Tablet
  Other Names: Marevan®
Drug: Omeprazole — 40 mg Tablet
  Other Names: Losec®; MUPS®
Drug: Midazolam — 5 mg/mL
  Other Names: Midazolam Accord®; versed
Drug: digoxin — .25 mg Tablet
  Other Names: lanoxin®
Drug: Vitamin K — 10 mg Tablet
  Other Names: warfarin antagonist
Drug: Rucaparib — 200 & 300 mg tablet
  Other Names: rucaparib camsylate; Rubraca; CO-338

SUMMARY:
The purpose of this study is to assess pharmacokinetic concentrations of multiple probes alone followed by assessment of the same drug pharmacokinetic concentrations when the patient has steady-state exposure to rucaparib followed by cycle-by-cycle treatment with rucaparib continuing until disease progression or other reason for discontinuation.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, sequential, drug-drug-interaction (DDI) study in patients with advanced solid tumors. The study will consist of 2 parts: a DDI part (Part I) and a rucaparib treatment part (Part II).

In Part I, the PK of cytochrome P450 (CYP) cocktail probes: caffeine, S-warfarin, omeprazole, and midazolam and a P-glycoprotein probe (digoxin) will be assessed with and without rucaparib treatment. Patients will receive single doses of CYP drug cocktail (caffeine, warfarin, omeprazole, and midazolam) on Day 1 and Day 12, and single doses of digoxin on Day 2 and Day 13. Continuous treatment with 600 mg rucaparib twice daily (BID) will start on Day 5 and will last until at least Day 16 of Part I.

In Part II, the treatment with rucaparib in 28-day cycles will continue until progression of disease, unacceptable toxicity, or other reason for discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced solid tumor
* Have evidence of measurable disease as defined by RECIST Version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate bone marrow, renal, and liver function

Exclusion Criteria:

* Prior treatment with chemotherapy, radiation, antibody therapy or other immunotherapy, gene therapy, vaccine therapy, angiogenesis inhibitors, or experimental drugs within 14 days prior to Day 1
* Prior treatment with any poly adenosine diphosphate ribose polymerase inhibitor (PARPi)
* Arterial or venous thrombi (including cerebrovascular accident), myocardial infarction, admission for unstable angina, cardiac angioplasty, stenting or poorly controlled hypertension within the last 3 months prior to Screening;
* Pre-existing duodenal stent, recent or existing bowel obstruction, and/or any gastrointestinal disorder or defect that would, in the opinion of the Investigator, interfere with absorption of study drugs
* Current use of therapeutic anticoagulation (low molecular weight heparin, oral anticoagulant agents including acetylsalicylic acid),
* Current use of one of the probe drugs;
* Untreated or symptomatic central nervous system (CNS) metastases.
* Evidence or history of bleeding disorder
* Participation in another investigational drug trial within 30 days prior to Day 1 (or 5 times the half-life of the drug, whichever is longer) or exposure to more than three new investigational agents within 12 months prior to Day 1;
* Acute illness within 14 days prior to Day 1 unless mild in severity and approved by the Investigator and Sponsor's medical representative
* Active second malignancy, i.e., patient known to have potentially fatal cancer present for which they may be (but not necessarily) currently receiving treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
PK parameters for caffeine, S-warfarin, omeprazole, midazolam, and digoxin with and without rucaparib treatment to be calculated from the plasma concentration-time data | Days 1-5 and Days 12-16
  Maximum plasma concentration [Cmax]
PK parameters for caffeine, S-warfarin, omeprazole, midazolam, and digoxin with and without rucaparib treatment to be calculated from the plasma concentration-time data | Days 1-5 and Days 12-16
  Area under the concentration-time curve (AUC) up to time t, where t is the last time point with concentrations above the lower limit of quantitation [AUC0-last ]

SECONDARY OUTCOMES:
PK parameters for caffeine, S-warfarin, omeprazole, midazolam, and digoxin with and without rucaparib treatment to be calculated from the plasma concentration-time data | Days 1-5 and Days 12-16
  Area Under the Curve, from time zero up to infinity with extrapolation of the terminal phase [AUC0-inf]
Tolerability and safety of rucaparib with and without co-administration of the probe drugs assessed by incidence of Adverse Events (AEs), clinical laboratory abnormalities, and dose modifications" | Days 1-16
  Incidence of Adverse Events (AEs), clinical laboratory abnormalities, and dose modifications
PK parameters will be calculated for rucaparib at steady-state | Day 7-12
  Trough plasma concentration [Ctrough]
PK parameters will be calculated for rucaparib at steady-state | Day 7-12
  Maximum plasma concentration during a dosing interval at steady-state [Cmax,ss]
PK parameters will be calculated for rucaparib at steady-state | Day 7-12
  Time to attain maximum plasma concentration at steady-state [tmax,ss]
PK parameters will be calculated for rucaparib at steady-state | Day 7-12
  Area Under the Curve over a dosing interval τ at steady-state [AUCτ,ss]
PK parameters for caffeine, S-warfarin, omeprazole, midazolam, and digoxin with and without rucaparib treatment to be calculated from the plasma concentration-time data | Days 1-5 and Days 12-16
  Terminal half-life [t1/2]
PK parameters for caffeine, S-warfarin, omeprazole, midazolam, and digoxin with and without rucaparib treatment to be calculated from the plasma concentration-time data | Days 1-5 and Days 12-16
  Time to attain maximum plasma concentration [tmax]
PK parameters for caffeine, S-warfarin, omeprazole, midazolam, and digoxin with and without rucaparib treatment to be calculated from the plasma concentration-time data | Days 1-5 and Days 12-16
  Apparent clearance [CL/F]
PK parameters for caffeine, S-warfarin, omeprazole, midazolam, and digoxin with and without rucaparib treatment to be calculated from the plasma concentration-time data | Days 1-5 and Days 12-16
  Apparent volume of distribution during terminal phase [Vz/F]

OTHER OUTCOMES:
Response will be determined using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 and tumor markers per applicable criteria for a given tumor type | From cycle 1 Day 1until radiologically confirmed disease progression, death, or initiation of subsequent treatment whichever comes first up to 52 weeks
  28 day cycles with response evaluation every 8 weeks(±7 days) until week 24 thereafter every 12 weeks (±14 days)

CONTACTS AND LOCATIONS:
Locations (3):
- Poland (3):
  - BioVirtus Research Site, Kajetany, Mokra 7
  - Med Polonia, Poznan
  - Zachodniopomorskie Centrum Onkologii Centrum Innowacji, Szczecin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xiao JJ, Nowak D, Ramlau R, Tomaszewska-Kiecana M, Wysocki PJ, Isaacson J, Beltman J, Nash E, Kaczanowski R, Arold G, Watkins S. Evaluation of Drug-Drug Interactions of Rucaparib and CYP1A2, CYP2C9, CYP2C19, CYP3A, and P-gp Substrates in Patients With an Advanced Solid Tumor. Clin Transl Sci. 2019 Jan;12(1):58-65. doi: 10.1111/cts.12600. Epub 2018 Dec 20. PMID 30427584